CLINICAL TRIAL: NCT04749472
Title: Biomechanical Analysis of Scapula and Humerus With Different Shoulder Slings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, assistant professor, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUSportsSling
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Shoulder Injuries; Surgery
Keywords: Rehabilitation; Shoulder Surgery; Postoperative
MeSH Terms: conditions — Shoulder Injuries | interventions — Suburethral Slings

STUDY DESIGN:
Intervention Model Description: Participants wore different sling in a randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Participants received intervention.
  Interventions: Other: Sling

INTERVENTIONS:
Other: Sling — Participants wore six different shoulder slings in a randomized order.

SUMMARY:
Participants will be measured with motion monitor system while using 6 different slings. Measurement order will be randomized, and 5 minutes resting period will be given prior measurement. Scapula, humerus and thorax positions will be recorded in resting position and then with slings.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Having a shoulder surgery
* Having scapular dyskinesis,
* Having shoulder pain,
* Having any disease that could affect posture and/or shoulder (such as scoliosis)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2022-09-12 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Motion Monitor | During rest position without and with different slings for 5 seconds.
  Motion monitor device was used to analyze 3D positions of the arm, shoulder, scapula and thorax.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)